CLINICAL TRIAL: NCT07292584
Title: Evaluating an Interactive Digital Toolkit for Women's PrEP Implementation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mirjam-Colette Kempf, University Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300015561; 000548592 (Other Grant/Funding Number: Gilead Sciences)
Record Dates: First submitted 2025-11-24; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: HIV Prevention; HIV Risk; Sexual and Reproductive Health
Keywords: PrEP; HIV prevention; cisgender women; Digital Health; Digital Intervention; Health Education; Decision Support Tool; Alabama; Mississippi; Southeast United States
MeSH Terms: conditions — Coitus; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation of interactive digital PrEP toolkit for increased PrEP uptake (Experimental): The goal of the intervention is to strengthen the PrEP care continuum by developing and testing an interactive digital PrEP toolkit designed to improve PrEP awareness, screening, engagement, retention, adherence, and persistence among individuals at increased risk for HIV seroconversion. Specifically, the intervention aims to reduce racial and gender disparities in PrEP uptake and use.
  Interventions: Behavioral: Interactive Digital PrEP Toolkit

INTERVENTIONS:
Behavioral: Interactive Digital PrEP Toolkit — Evaluation of an Interactive Digital PrEP Toolkit for women in AL and MS

SUMMARY:
The goal of this study is to test if a Digital PrEP Toolkit helps cisgender women learn about and access PrEP in Alabama and Mississippi. PrEP is a medication that prevents HIV infection. The main questions it aims to answer are: Can participants complete the Digital PrEP Toolkit in under 10 minutes? Do participants find the Digital PrEP Toolkit useful and easy to use? Does the Digital PrEP Toolkit increase the number of women who start taking PrEP?

Investigators will work with up to 125 women at 3 HIV and STI clinics in Alabama and Mississippi.

Participants will use the Digital PrEP Toolkit on a tablet at the clinic. They will answer questions about their HIV knowledge before and after using the Toolkit. Participants will then discuss PrEP options with a healthcare staff member and decide if they want to start PrEP. Participants will answer follow-up questions at 3 months. Investigators will also review participants' medical records at 6 months to see if they started PrEP and are still taking it.

DETAILED DESCRIPTION:
Cisgender women in the rural southeastern United States face substantial HIV risk. Despite this, pre-exposure prophylaxis (PrEP) use among women remains alarmingly low. PrEP is a medication that prevents HIV infection. Barriers to PrEP use among women include limited PrEP awareness and knowledge, low HIV risk perception, challenging client-provider conversations about sexual health, and structural challenges like transportation difficulties and time constraints.

This study will test an Interactive Digital PrEP Toolkit that includes HIV prevention education tailored to women in the Southeast, information about different PrEP medication options (i.e., daily oral pills, monthly injections, and twice-yearly injections), questions to help identify HIV prevention preferences, and testimonials from women using PrEP. The study will enroll up to 125 cisgender women at 3 HIV and STI clinic locations in Alabama and Mississippi over approximately 12 months.

Study Outcomes:

Primary outcomes include feasibility, acceptability, and preliminary efficacy. Feasibility will be measured by Toolkit completion rate, average time to complete the Toolkit, proportion of participants who initiate PrEP, and changes in HIV and PrEP knowledge. Acceptability will be measured through participant satisfaction surveys assessing how valuable and easy to use participants find the Digital PrEP Toolkit. Preliminary efficacy will be measured by comparing clinic-level PrEP uptake rates during up to 12 months preceding the study start to those during the approximately 12-month study period among all eligible female clients seen at participating clinics.

Secondary outcomes will include documentation of participants' sexual health priorities, HIV prevention preferences, and PrEP modality choices across the clinic sites. Investigators will also assess retention in PrEP care at 6 months post-enrollment.

Study Procedures:

Participants will complete a 30-minute enrollment visit at the clinic. They will provide informed consent, complete baseline assessments on HIV and PrEP knowledge, health-related questions, and demographics, and use the Interactive Digital PrEP Toolkit on a tablet. After completing the Toolkit, participants will receive a Personalized HIV Prevention Summary and meet with a healthcare staff member to discuss PrEP. Participants interested in PrEP will be scheduled for a PrEP clinic appointment.

At 3 months, Research staff will contact participants by phone for a follow-up interview about HIV and PrEP knowledge, sexual health, PrEP uptake and adherence, and experiences with the Toolkit. Research staff will also review medical records at 3 months for PrEP prescriptions.

At 6 months, research staff will review medical records for continued PrEP prescriptions. Participants will not be contacted at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative
* Cisgender women
* 18 years or older
* English-speaking
* Report sexual activity in the last six months or anticipate sexual activity in the next six months.

Exclusion Criteria:

* Younger than 18 years of age
* Do not identify as female and/or were not biologically assigned female at birth
* Living with HIV
* Report no sexual activity in the past six months and no anticipated sexual activity in the next six months
* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 125 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Toolkit completion rate | Throughout 12-month enrollment period
  Percentage of eligible women who complete the PrEP Toolkit out of women screened and enrolled
Feasibility: Toolkit Completion Time | Throughout 12-month enrollment period
  Average time needed to complete PrEP Toolkit activities
Acceptability: Participant Satisfaction | From enrollment to the end of the 3 month follow-up period at 15-months
  Participant satisfaction will be assessed using a study-specific satisfaction questionnaire measuring perceived value and ease of use of the Digital PrEP Toolkit. The questionnaire includes Likert-scale items (range: 1-5, with higher scores indicating greater satisfaction) evaluating Toolkit usability, perceived usefulness, and overall satisfaction.
Preliminary Efficacy: Participant PrEP Uptake | From enrollment to the end of the 3 month follow up period at 15-months
  Proportion of eligible women who initiate PrEP after using the PrEP Toolkit to eligible clients screened
Preliminary Efficacy: Clinic-level PrEP uptake | From enrollment to the end of the 3 month follow up period at 15-months
  Comparison of PrEP uptake rates up to 12-months prior to study start to PrEP uptake rates during the approximately 12-month study enrollment period among eligible women at the partnering clinic sites
Preliminary Efficacy: HIV and PrEP Knowledge | From enrollment to the end of the 3 month follow up period at 15-months
  Changes in HIV and PrEP knowledge will be assessed using an adapted version of the updated HIV Knowledge Questionnaire (range: 0-31, with higher scores indicating greater knowledge).

SECONDARY OUTCOMES:
Number of Participants by Sexual Health Priority | Throughout 12-month enrollment period
  Documentation of participants' sexual health priorities will be assessed using a study-specific questionnaire capturing: (1) reasons for PrEP consideration, and (2) factors most important to participants when considering HIV prevention and sexual wellness (e.g., effectiveness, convenience, privacy, cost).
Number of Participants by HIV Prevention Preference | Throughout 12-month enrollment period
  Participants' HIV prevention preferences will be assessed using a study-specific questionnaire capturing stated interest in daily PrEP, injectable PrEP, both options, non-medication options, or no current interest.
Number of Participants by PrEP Modality Choice | From enrollment to the end of the 3 month follow up period at 15-months
  Documentation of clients' decisions on PrEP methods (e.g., oral, injectable)
PrEP Persistence | From enrollment to the end of the 6 month follow up period at 18-months
  Proportion of clients who initiated PrEP and continue to be engaged in PrEP care at 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam-Colette Kempf, PhD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Five Horizons Health Services, Montgomery, Alabama
  - Five Horizons Health Services, Tuscaloosa, Alabama
  - Five Horizons Health Services, Starkville, Mississippi

IPD SHARING:
Plan to Share IPD: Yes
Our current plans call for the results of the process and outcome evaluations collected as part of this project will be shared via professional presentations and publications and will also be shared upon request. De-identified data will also be electronically encrypted and archived for use by others who are interested in using this data. New procedures, protocols, data collection instruments and analytic routines will be made available to interested investigators.
Time Frame: Data will be available after analysis is completed.
Access Criteria: Only de-identified information will be available.